CLINICAL TRIAL: NCT04139252
Title: A National Study for Blood Based Response Monitoring of Newly Diagnosed Aggressive B-cell Lymphoma (DLBCL and HGBCL) Patients
Brief Title: A National Study for Blood Based Response Monitoring of B-cell Lymphoma Patients
Acronym: HO902DLBCL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Other Study IDs: HO902
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: NHL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Observational prospective study. Patients with DLBCL and HGBCL will be enrolled in the study to collect samples for developing a blood based assay allowing biomarker driven treatment in the future.

DETAILED DESCRIPTION:
The rationale of this study is that, due to the lack of successful salvage options, first-line treatment outcome needs to be improved. To make this possible, a crucial condition is optimal identification of patients that will not be cured on R-CHOP. The aim of this protocol is to develop new tools to monitor treatment response and disease outcome. Molecular monitoring of treatment response through liquid biopsies (LB) is such a promising new tool.

The primary objective is to collect liquid biopsy samples of patients with newly diagnosed DLBCL/HGBCL to develop a blood based assay allowing biomarker driven treatment in the future.

The secondary objectives are to collect clinical data and pre-treatment tissue samples (for determining molecular profiles) to allow for correlation to the blood based assay.

This study is designed for patients with newly diagnosed DLBCL and HGBCL ≥ 18 yr.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with newly diagnosed DLBCL (including HGBCL- NOS and HGBCL-DH) according to WHO classification 2016
* Ann Arbor stage II-IV
* Patients intended to be treated with 6 cycles R-CHOP (or DA-EPOCH-R) as first-line treatment (successive inclusion in HOVON 151 or HOVON 152 is possible)
* Age ≥ 18 years

Exclusion Criteria:

- Patients with limited stage I, II disease planned to receive 3 cycles of R-CHOP + radiotherapy, or 4 x R-CHOP+ 2R

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Tissue material | 24 months
  For genomic analysis and clinical outcome data

CONTACTS AND LOCATIONS:
Overall Officials: M.E.D. Chamuleau, MD, PhD, Principal Investigator — VUmc
Locations (60):
- Netherlands (60):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Alkmaar-NWZ, Alkmaar
  - NL-Almelo-ZGTALMELO, Almelo
  - NL-Almere-FLEVOZIEKENHUIS, Almere Stad
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amstelveen-AMSTELLAND, Amstelveen
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Assen-WZA, Assen
  - NL-Beverwijk-RKZ, Beverwijk
  - NL-Breda-AMPHIA, Breda
  - NL-Capelle a/d IJssel-YSL, Capelle aan den IJssel
  - NL-Delft-RDGG, Delft
  - NL-Deventer-DZ, Deventer
  - NL-Dirksland-VANWEELBETHESDA, Dirksland
  - NL-Doetinchem-SLINGELAND, Doetinchem
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Ede-ZGV, Ede
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Emmen-SCHEPER, Emmen
  - NL-Enschede-MST, Enschede
  - NL-Geldrop-STANNA, Geldrop
  - NL-Goes-ADRZ, Goes
  - NL-Gorinchem-BEATRIX, Gorinchem
  - NL-Gouda-GROENEHART, Gouda
  - NL-Groningen-UMCG, Groningen
  - NL-Hardenberg-SAXENBURGH, Hardenberg
  - NL-Harderwijk-STJANSDALHARDERWIJK, Harderwijk
  - NL-Heerenveen-TJONGERSCHANS, Heerenveen
  - NL-Helmond-ELKERLIEK, Helmond
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Hoorn-DIJKLANDERHOORN, Hoorn
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Roermond-LZR, Roermond
  - NL-Roosendaal-BRAVIS, Roosendaal
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Rotterdam-IKAZIA, Rotterdam
  - NL-Rotterdam-MAASSTADZIEKENHUIS, Rotterdam
  - NL-Rotterdam-SFG, Rotterdam
  - NL-Sneek-ANTONIUSSNEEK, Sneek
  - NL-Spijkenisse-SPIJKENISSEMC, Spijkenisse
  - NL-Terneuzen-ZORGSAAM, Terneuzen
  - NL-Den Haag-HAGA, The Hague
  - NL-Den Haag-HMCWESTEINDE, The Hague
  - NL-Tiel-RIVIERENLAND, Tiel
  - NL-Tilburg-ETZ, Tilburg
  - NL-Uden-BERNHOVEN, Uden
  - NL-Utrecht-DIAKONESSENUTRECHT, Utrecht
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Venlo-VIECURI, Venlo
  - NL-Winterswijk-SKBWINTERSWIJK, Winterswijk
  - NL-Zutphen-GELREZUTPHEN, Zutphen
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: No